CLINICAL TRIAL: NCT06218758
Title: Prediction Model for Postoperative Pulmonary Complications in Patients Undergoing Lung Transplantation Using Machine Learning: a Retrospective Cohort Study
Brief Title: Prediction Model for PPCs in Patients Undergoing Lung Transplantation Using Machine Learning
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Assistant professor for fund, Pusan National University Yangsan Hospital
Other Study IDs: 55-2024-004
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplantation
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: General anesthesia — General anesthesia using 2% propofol, and remifentanil for lung transplantation

SUMMARY:
Since the first human lung transplantation in 1963, significant advancements in immunosuppressive agents from the mid-1990s have greatly improved the quantity and quality of such procedures. In 2004, a total of 1,815 lung transplantations were globally reported. Patients undergoing this procedure are typically elderly and experience not only impaired lung function but also overall health instability. Despite successful outcomes, postoperative pulmonary complications (PPCs) can lead to serious consequences, including deterioration and fatality. PPCs resulting from lung transplantation may lead to prolonged hospitalization, increased complications, and the need for additional treatment. Various factors, such as age, smoking, pre-existing lung diseases, immunosuppressive drug use, diabetes, hypertension, infections, allergies, and immune disorders, are associated with the development of PPCs. The retrospective analysis of medical records from adult patients who underwent lung transplantation aims to investigate patient characteristics, anesthesia methods, intraoperative tests, and the occurrence of PPCs, with the ultimate goal of analyzing the incidence and risk factors of postoperative respiratory complications and developing a predictive model through machine learning.

DETAILED DESCRIPTION:
After the first report of lung transplantation in humans in 1963, rapid advancements in immunosuppressive agents since the mid-1990s have led to significant progress in both the quantity and quality of lung transplantation. In 2004, a total of 1,815 lung transplantations were reported worldwide. Patients undergoing lung transplantation are typically elderly, often experiencing not only impaired lung function but also overall instability in their health. Despite successful outcomes in lung transplantation, the occurrence of pulmonary complications after surgery can lead to deterioration or even fatal consequences.

Postoperative pulmonary complications (PPCs) can result in prolonged hospitalization, increased complications, and the need for additional treatment. Various factors are associated with the development of PPCs after lung transplantation, including age, smoking, pre-existing lung diseases (such as chronic obstructive pulmonary disease, pulmonary fibrosis, etc.), immunosuppressive drug use post-transplant, diabetes, hypertension, pulmonary hypertension, heart disease, infections, allergies, and immune disorders. The retrospective analysis of medical records of adult patients who underwent lung transplantation aims to investigate patient characteristics, anesthesia methods, intraoperative tests, and the occurrence of PPCs. The goal is to analyze the incidence and risk factors of postoperative respiratory complications and develop a predictive model through machine learning.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older who underwent lung transplantation for end-stage lung disease

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 years of age or older who underwent lung transplantation for end-stage lung disease
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | Up to 1 year after lung transplantation
  Postoperative pulmonary complications such as pleural effusion, pneumothorax, hemothorax, chylothorax, atelectasis, pulmonary edema, acute respiratory distress syndrome, pneumonia, bronchial stenosis, pulmonary fibrosis and emphysema, postoperative tracheostomy, acute rejection occurring within the first year after lung transplantation, chronic rejection

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Department of Anesthesia and Pain Medicine, School of Medicine, Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No